CLINICAL TRIAL: NCT01705093
Title: The Effects of California Strawberries on Parameters of Cardiovascular Health
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 333071
Record Dates: First submitted 2012-08-31; First posted 2012-10-12 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Childhood Obesity; Cardiovascular Disease
Keywords: strawberry, cardiovascular, obesity, adolescent
MeSH Terms: conditions — Pediatric Obesity; Cardiovascular Diseases; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flavonoid-rich freeze-dried strawberry powder (Experimental): 50g of flavonoid-rich freeze-dried strawberry powder
  Interventions: Dietary Supplement: flavonoid-rich freeze-dried strawberry powder
- macronutrient- matched control powder (Placebo Comparator): 50g macronutrient-matched control powder that will lack strawberry flavonoids
  Interventions: Dietary Supplement: macronutrient-matched control powder

INTERVENTIONS:
Dietary Supplement: flavonoid-rich freeze-dried strawberry powder — 50g of flavonoid-rich freeze-dried strawberry powder
  Arms: Flavonoid-rich freeze-dried strawberry powder
Dietary Supplement: macronutrient-matched control powder — 50g macronutrient-matched powder that will lack strawberry flavonoids
  Arms: macronutrient- matched control powder

SUMMARY:
The prevalence of childhood obesity has been increasing over the past couple of decades. Similar to adults, overweight and obesity in young children and adolescents is associated with an increased number of cardiovascular risk factors including dyslipidemia, hypertension, insulin resistance and Type 2 diabetes. Epidemiological and clinical studies suggest that foods and ingredients rich in select flavonoids, such as cocoa, red grape products, tea, citrus fruits, and strawberries are protective against the development of cardiovascular disease. Strawberries are rich in flavonoids, particularly anthocyanins, flavanols, flavonols, ellagic acid and its glucose ester, ellagitanin. A number of in vitro studies have observed that these isolated compounds, as well as strawberry extracts have the potential to affect outcomes of cardiovascular health, including vascular reactivity, cellular signaling and oxidant defense6,7. We hypothesize that strawberry intake will lead to improvements in select measures of cardiovascular function in overweight and obese adolescent males.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, age 14 - 18 years.
* BMI for age and gender >75th percentile (based on CDC growth charts)
* Subject is willing and able to comply with the study protocols.

Exclusion Criteria:

* Inability to wear PAT probes
* Inability to remain still and remain quiet during test procedures
* BMI for age and gender ≤ 75th percentile (based on CDC growth charts)
* The use of medications that affect vascular function
* Regular use of dietary supplements during the last 6 months
* Blood pressure for age, gender and height ≥95th percentile
* Chronic/routine high intensity exercise or current participation in a sports program
* Self/Parent reported use of anticoagulation agents including NSAIDs
* Self/Parent reported use of oral cortisone or other immunosuppressive agents,
* Self/Parent reported underlying neoplasia or immunological disease
* Self/Parent reported diabetes
* Food faddists or those taking a non-traditional diet
* Allergies to fruit
* Abnormal Liver, CBC or Chemistry panels (laboratory values outside the reference
* range) if determined to be clinically significant by the study physician.
* Self/Parent reported malabsorption (e.g. difficulty digesting or absorbing nutrients from food, potentially leading to bloating, cramping or gas).
* Asthma (can be worsened by mild to moderate food allergies).

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Vascular function measured by peripheral arterial tonometry | Change from baseline in vascular function at 1 hour and 1 week
  Change from baseline at 1 hour and 1 week post consumption of freeze-dried strawberry powder or control powder

CONTACTS AND LOCATIONS:
Locations (1):
- Ragle Human Nutrition Research Center, Academic Surge, UC Davis, Davis, California, United States